CLINICAL TRIAL: NCT01513265
Title: Rationalisation of Polypharmacy in the Elderly by the RASP Instrument (Rationalisation of Home Medication by an Adjusted STOPP-list in Older Patients): a Prospective, Clinical Trial.
Brief Title: Rationalisation of Polypharmacy in the Elderly by the RASP Instrument
Acronym: RASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S-53664
Record Dates: First submitted 2011-12-27; First posted 2012-01-20 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: reduction polypharmacy; clinical outcomes; pharmaceutical care; clinical pharmacy; geriatrics; medication review; potentially inappropriate drugs

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- RASP (Active Comparator)
  Interventions: Other: Pharmaceutical care plan, mostly based on the RASP
- Control group (No Intervention): Subjects enrolled in this arm will undergo usual medical and pharmaceutical care with registration of drug use at admission and discharge without interference of RASP or clinical pharmacist.

INTERVENTIONS:
Other: Pharmaceutical care plan, mostly based on the RASP — Drug use of subjects enrolled in this arm will be systematically evaluated by a clinical pharmacist, using the RASP list. Potentially inappropriate drug use will be pointed out to the treating physician. The pharmaceutical advice is not limited to the RASP list. Any actual change in drug prescription will be decided by the treating physician based upon comprehensive medical evaluations in each individual patient.
  Arms: RASP

SUMMARY:
The aim of this study is to determine whether a clinical pharmacist using the RASP list (RASP = Rationalisation of home medication by an adjusted STOPP-list in older patients; STOPP = Screening Tool of Older Persons' potentially inappropriate Prescriptions) can optimise the drug use in elderly inpatients.

DETAILED DESCRIPTION:
Older persons take on average multiple drugs. As people age, there is an apparent increase in pharmacodynamic sensitivity to different making the patient more prone to experience side effects. Alterations in body composition and concomitant changes in pharmacokinetic parameters can also result in a higher risk for adverse drug events. All these factors make the older person, notwithstanding the heterogeneity of this population, more vulnerable for the negative consequences of polypharmacy.

Polypharmacy is a cause of negative clinical outcomes but it still remains unclear which intervention or set of interventions should be used to optimize the prescription of pharmacotherapy in the elderly patient. Therefore, the investigators developed the RASP (RASP = Rationalisation of home medication by an adjusted STOPP-list in older patients; STOPP = Screening Tool of Older Persons' potentially inappropriate Prescriptions), a list as tool to reduce polypharmacy adapted to Belgian national prescribing tendencies within geriatric wards. Content and reliability of the RASP have been validated and the investigators aim to further study the impact of the systematic implementation of this RASP on geriatric wards in a prospective cluster randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the patient or a caregiver if the patient is incompetent to sign
* Consecutive inclusion of all newly admitted patients to the wards coming from home or the emergency room department

Exclusion Criteria:

* Patients not admitted to the hospital from home or a nursing home
* Patients unable to communicate in Dutch
* Patients admitted for palliative care
* Patients who do not take any drugs at admission

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of actually stopped or adjusted drugs | Patients will be followed for the duration of hospital stay, an expected average of 14 days.
  At hospital discharge the number of stopped or adjusted drugs will be determined. This variable will be compared between the two arms.

SECONDARY OUTCOMES:
Number of potentially inappropriate drug prescriptions as defined by the RASP. | Patients will be followed for the duration of hospital stay, an expected average of 14 days.
Actual drug use | Measured on 30 and 90 days post-discharge.
Number and category of drugs adjusted on recommendations of the clinical pharmacist independent of RASP | Patients will be followed for the duration of hospital stay, an expected average of 14 days.
Mortality | Measured during hospitalisation, an expected average of 14 days and within 90 days after discharge.
Number of falls | Measured during hospitalisation, an expected average of 14 days and within 90 days after discharge
Quality of Life (EQ-5D-3L) | Patients will be followed for the duration of hospital stay, an expected average of 14 days.
Length of stay | Determined at discharge, on average after 14 days
Rehospitalisation | Within 90 days post-discharge.
Incidence of delirium | Patients will be followed for the duration of hospital stay, an expected average of 14 days
Number of falls post-discharge | Within 90 days post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Van der Linden, PharmD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Van der Linden L, Decoutere L, Walgraeve K, Milisen K, Flamaing J, Spriet I, Tournoy J. Combined Use of the Rationalization of Home Medication by an Adjusted STOPP in Older Patients (RASP) List and a Pharmacist-Led Medication Review in Very Old Inpatients: Impact on Quality of Prescribing and Clinical Outcome. Drugs Aging. 2017 Feb;34(2):123-133. doi: 10.1007/s40266-016-0424-8. PMID 27915457